CLINICAL TRIAL: NCT01361178
Title: Immunoglobulin Levels and Occurrence of Infections After Lung Transplantation and Impact of IgG Replacement - Observational Arm
Brief Title: Immunoglobulin Levels and Occurrence of Infections After Lung Transplantation and Impact of IgG Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Andrej Petrov, Andrej Petrov, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09090483
Record Dates: First submitted 2011-05-13; First posted 2011-05-26 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Infections After Lung Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant patients who do not receive SQ IVIG (No Intervention): Patients participating in the observational arm of the study who do not need to receive IgG replacement.
- Transplant patients who receive SQ IVIG (Active Comparator): Patients participating in the observational arm of the study who are randomized to receive a dosage of SQ IVIG due to low IgG level.
  Interventions: Drug: SQ IVIG

INTERVENTIONS:
Drug: SQ IVIG — Group 1 will receive SQ IgG at the lower end of the dosing range at 100 mg/kg/week and group 2 will receive SQ IgG at the higher end of the dosing range at 200 mg/kg/week
  Arms: Transplant patients who receive SQ IVIG

SUMMARY:
Immunosuppressive therapies have led to remarkable improvements in survival in lung transplantation (LT) patients. However, one important adverse effect of these therapies has been the increasing emergence of hypogammaglobulinemia (HGG) which has been previously seen mostly in patients with primary immunodeficiency (PID).

The goal of treatment of HGG in PID has been to maintain the trough IgG level above 500 mg/dl which might provide better protection against infections than do lower IgG serum concentrations. Although IgG therapy is of substantial benefit, the doses and trough levels of IgG that are optimal are not yet clearly established. The impact of high versus low IgG dosing on the frequency and severity of infections and rejection has not been studied before in LT patients with HGG. The specific aims for this study are to compare the incidence of infections in lung transplant recipients receiving higher versus lower dose of SQ IgG and to compare the incidence of infections in lung transplant recipients with mild hypogammaglobulinemia versus normal IgG levels. This study will be a single center study of all lung transplant recipients, age 18 years or older, at the University of Pittsburgh Medical Center (UPMC), with a randomized treatment arm and an observational arm.

The hypotheses for the research study are:

* Therapy with IV or SQ IgG is of substantial benefit in reducing the number of infections in lung transplant recipients with severe hypogammaglobulinemia (IgG < 500)
* A higher dose of SQ IgG, with subsequent higher trough IgG levels, may have a higher impact on the frequency and severity of infections and rejection episodes, compared to a lower dose of SQ IgG, with subsequent lower IgG trough levels
* Lung transplant recipients with mild hypogammaglobulinemia ( IgG= 500-750) have a higher incidence of infections compared to patients with normal IgG levels

ELIGIBILITY:
Inclusion Criteria:

* adult recipients of lung transplantation at the University of Pittsburgh Medical Center, who are able to provide written informed consent prior to transplantation or on the day of lung transplant surgery.

Exclusion Criteria:

* age less than 18 years-old
* history of anaphylaxis to IVIG
* subjects already on IV or SQ IgG treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Comprehensive Lung Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transplant Patients Who do Not Receive SQ IVIG | Transplant Patients Who Receive SQ IVIG
Started | 122 | 11
Completed | 109 | 11
Not Completed | 13 | 0
Not completed — Death | 13 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transplant Patients Who do Not Receive SQ IVIG | Transplant Patients Who Receive SQ IVIG | Total
Number analyzed (Participants) | 122 | 11 | 133
Age, Continuous [Median (Full Range); unit: years] | 62 [18 to 75] | 52 [26 to 70] | 61 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 5 | 51
  Male | 76 | 6 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 113 | 11 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Diagnosis [Count of Participants; unit: Participants]
  IPF | 44 | 2 | 46
  COPD | 37 | 3 | 40
  Cystic Fibrosis | 10 | 3 | 13
  Scleroderma | 11 | 1 | 12
  Sarcoidosis | 3 | 1 | 4
  Pulmonary Hypertension | 3 | 0 | 3
  Other | 14 | 1 | 15
Induction Agent [Count of Participants; unit: Participants]
  Alemtuzamab | 84 | 5 | 89
  Basiliximab | 38 | 6 | 44

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Will be the Total Number of Days With Pneumonia.
Description: The primary outcome for this study will be the total number of days with pneumonia. Pneumonia will be defined by the presence of both clinical and radiographic criteria: fever (temperature ≥ 38oC), cough, dyspnea, purulent expectoration and/or changes in the previous characteristics of respiratory secretions; and chest X-ray or CT scan revealing a new or progressive alveolar or interstitial infiltrate or cavitation that could not be explained by any other noninfectious cause.
Time Frame: Up to two years post-transplant
Measure: Number; unit: Number of days
Arm/Group | Transplant Patients Who do Not Receive SQ IVIG | Transplant Patients Who Receive SQ IVIG
Number analyzed (Participants) | 122 | 11
Number of days | 1714 | 51

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Transplant Patients Who do Not Receive SQ IVIG | Transplant Patients Who Receive SQ IVIG
All-Cause Mortality (participants affected / at risk) | 13/122 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/11
Other Adverse Events (participants affected / at risk) | 0/122 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes